CLINICAL TRIAL: NCT01728857
Title: The Effects of Tissue Optimization on Cryolipolysis Procedures for Fat Layer Reduction
Brief Title: Tissue Optimization on Cryolipolysis Procedures for Fat Layer Reduction
Acronym: TOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA12-007
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Body Fat Disorder
Keywords: Lipolysis; Cryolipolysis; Fat Reduction
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fat Reduction (Experimental)
  Interventions: Device: The Zeltiq System

INTERVENTIONS:
Device: The Zeltiq System — Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
  Other Names: Cryolipolysis; Lipolysis

SUMMARY:
Evaluate the effects of tissue optimization before and during cryolipolysis procedures on the outcome of non-invasive fat reduction using the ZELTIQ System.

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects > 18 years of age and < 65 years of age.
2. Subject has clearly visible fat on intended treatment area, which in the investigator's opinion, may benefit from the treatment(s).
3. Subject has not had weight change exceeding 10 pounds in the preceding month.
4. Subject with body mass index (BMI) less than 30. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
5. Subject agrees to maintain his/her weight (i.e., within 5 pounds) by not making any major changes in their diet or lifestyle during the course of the study.
6. Subject has read and signed a written informed consent form.

Exclusion Criteria

1. Subject presents a significant asymmetry of intended treatment areas.
2. Subject has had a surgical procedure(s) in the area of intended treatment in the past 5 years.
3. Subject has had an invasive fat reduction procedure (e.g., liposuction, abdominoplasty, mesotherapy) in the area of intended treatment in the past 5 years.
4. Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 6 months.
5. Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
6. Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
7. Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
8. Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
9. Subject is taking or has taken diet pills or weight control supplements within the past month.
10. Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
11. Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system.
12. Subject is pregnant or intending to become pregnant in the next 5 months.
13. Subject is lactating or has been lactating in the past 6 months.
14. Subject has a history of hernia in the areas to be treated.
15. Subject is unable or unwilling to comply with the study requirements.
16. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
17. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2014-03-10 (Actual); Study Completion 2014-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Development - Body Contouring, Study Director — Zeltiq Aesthetics
Locations (1):
- Innovation Research Center, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who consented to participate in the study underwent a screening period of 90 days.
Groups:
- The ZELTIQ System: Participants received cryolipolysis treatment in the abdomen area for fat layer reduction on Day 0.
Period: Overall Study
Arm/Group | The ZELTIQ System
Started | 19
Received at Least 1 Study Treatment | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received the study treatment.
Arm/Group | The ZELTIQ System
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 41.4 [27.2 to 56.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Before and After Side-by-side Photographs Correctly Identified by At Least 2 of 3 Blinded Reviewers From the Independent Physician Reviewer (IPR) Panel
Description: Photographs of the treatment areas were taken at baseline, and at 16-weeks after the first treatment with the ZELTIQ System were assessed for any visual changes. The photographs were assessed by blinded independent reviewers (IPR) to correctly identify the 16-weeks post-treatment photographs from randomly placed side-by-side comparison of before and after photographs. Reported here is the percentage (%) of images that were correctly identified by at least 2 out of 3 blinded independent reviewers.
Time Frame: Baseline, Week 16
Population: Per-protocol Population included all the treated participants followed for 16 weeks post-treatment with weight change of no more than five pounds at the Week 16 visit.
  Here, 'Overall Number of Participants Analyzed' is the number of participants evaluable for this Endpoint.
Measure: Number (95% Confidence Interval); unit: % of images identified correctly
Units Other Than Participants: images
Arm/Group | The ZELTIQ System
Number analyzed (Participants) | 13
Number analyzed (images) | 13
% of images identified correctly | 30.8 [9.1 to 61.4]

2. Secondary Outcome: Change From Baseline in Reduction of Fat Layer Thickness as Assessed by Ultrasound
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | The ZELTIQ System
Number analyzed (Participants) | 13
centimeters (cm) | -0.14 (0.21)

ADVERSE EVENTS:
Time Frame: From date of first treatment up to Week 16
Description: Safety Population included all participants who received the study treatment, with available safety evaluation after the treatment.
Arm/Group | The ZELTIQ System
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 5/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | The ZELTIQ System (N=19)
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Stool impaction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Common Cold/Respiratory Infection (General disorders) | 1
Cough (General disorders) | 1
Nasal congestion (General disorders) | 1
Sore throat (General disorders) | 1
Firmness or discrete nodules within the treatment area (Musculoskeletal and connective tissue disorders) | 1
Numbness, tingling, burning lasting longer than 8 weeks (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Zeltiq requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Zeltiq requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Zeltiq needs to secure patent or proprietary protection.